CLINICAL TRIAL: NCT05299125
Title: A Single Arm, Phase 2 Study of Amivantamab, Lazertinib and Pemetrexed for First-line Treatment of Recurrent/Metastatic Non-small Cell Lung Cancers (NSCLCs) With EGFR Mutations
Brief Title: Amivantamab, Lazertinib, and Pemetrexed for First-line Treatment of Recurrent/Metastatic Non-small Cell Lung Cancers With Epidermal Growth Factor Receptor Mutations
Acronym: AMIGO-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0821; 73841937LUC2002 (Other Grant/Funding Number: Janssen)
Record Dates: First submitted 2022-02-25; First posted 2022-03-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Non-small Cell Lung Cancers
MeSH Terms: interventions — amivantamab; lazertinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Therapy consisting of lazertinib plus amivantamab plus chemotherapy (Experimental): CYCLE 1 (21-day cycle) Amivantamab 1400 mg (1750 mg if body weight is >80 kg) IV once weekly + Lazertinib 240 mg po daily + Pemetrexed 500 mg/m² IV on day 1
  CYCLE 2 (21-day cycle) Amivantamab 1400 mg (1750 mg if body weight is >80 kg) IV on day 1 + Lazertinib 240 mg po daily + Pemetrexed 500 mg/m² IV on day 1
  MAINTENANCE CYCLES 3 - 8 (21-day cycle) Amivantamab 1750 mg (2100 mg if body weight is >80 kg) IV on day 1 + Lazertinib 240 mg po daily + Pemetrexed 500 mg/m² IV on day 1
  MAINTENANCE CYCLES 9 + (21-day cycle) Amivantamab 1750 mg (2100 mg if body weight is >80 kg) IV on day 1 + Lazertinib 240 mg po daily
  Interventions: Drug: Amivantamab; Drug: Lazertinib; Drug: Pemetrexed 500 mg

INTERVENTIONS:
Drug: Amivantamab — Low fucose, fully human immunoglobulin gamma-1-based bispecific antibody directed against EGFR and MET tyrosine kinase receptors. It shows clinical activity against tumors with the primary activating EGFR mutations Exon 19del or Exon 21 L858R substitution, EGFR Exon 20ins mutations, the EGFR resistance mutations Threonine790Methionine (T790M) or Cysteine797Serine (C797S), and activation of the Mesenchymal Epithelial Transition (MET) pathway.
Drug: Lazertinib — It selectively inhibits both primary activating EGFR mutations (Exon 19del, Exon 21 L858R substitution) and the EGFR T790M resistance mutation, while having less activity versus wild-type EGFR.
Drug: Pemetrexed 500 mg — Inhibits enzymes involved in folate-dependent metabolism, thereby disrupting cellular replication.

SUMMARY:
This is a phase II, single-arm, multicenter trial, conducted through Latin American Coorperative Oncology Group (LACOG). Treatment-naïve patients with recurrent/metastatic NSCLCs harboring EGFR exon 19 deletions or exon 21 L858R point mutations will be enrolled. At baseline, an archival or (optional) new tissue sample will be obtained for biomarker evaluation, as well as liquid biopsies. Treatment will continue until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
This study aims to test the hypothesis that delivery of maximum therapy consisting of lazertinib plus amivantamab plus chemotherapy as frontline treatment in patients with recurrent/metastatic NSCLC with EGFR exon 19 or exon 21 mutations will be feasible, safe, and will improve PFS compared to historical controls. If successful, this study may allow for the estimation of efficacy and toxicity of a three drug regimen of amivantamab, lazertinib, and pemetrexed and may support further evaluation of maximum therapy against osimertinib single agent, lazertinib single agent, osimertinib plus chemotherapy, and/or lazertinib plus amivantamab.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age;
2. Participant must have histologically or cytologically confirmed locally advanced or metastatic NSCLC not amenable to curative therapy. Participants must be treatment-naïve for metastatic NSCLC. Prior adjuvant and neo-adjuvant therapy for early-stage disease is permitted, prior systemic therapy for potentially curable locally advanced disease is also permitted;
3. Participant must have a tumor that was previously determined to have Exon 19del or Exon 21 L858R substitution, as detected by a validated test in accordance with site standard of care. Note: A copy of the test report documenting the EGFR mutation must be included in the participant records and must also be submitted to the sponsor prior to enrollment;
4. Unstained tumor tissue and blood (for ctDNA, biomarker), both collected prior to treatment initiation, must be provided. Unstained FFPE tumor tissue blocks must be provided whenever possible. Alternatively, re-cut unstained sections from FFPE tumor tissue block, presented on slides must be provided (recommended 10-15 slides);
5. Subject must have specific organ and bone marrow function;
6. Participant must have ECOG status of 0 to 2;
7. Any toxicities from prior anticancer therapy must have resolved to CTCAE Grade 1 or baseline level;
8. Participant must have at least 1 measurable lesion, according to RECIST v1.1 that has not been previously irradiated. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

Exclusion Criteria:

1. Participant has received any prior systemic treatment for metastatic disease (prior systemic therapy for potentially curable locally advanced disease, adjuvant or neoadjuvant therapy are allowed, if administered more than 12 months prior to the development of the recurrent disease);
2. Participant has symptomatic brain metastases. A participant with asymptomatic or previously treated and stable brain metastases may participate in this study. Participants who have received definitive radiation or surgical treatment for symptomatic or unstable brain metastases and have been clinically stable and asymptomatic for at least 2 weeks before Screening are eligible, provided they have been either off corticosteroid treatment or are receiving low-dose corticosteroid treatment (≤10 mg/day prednisone or equivalent) for at least 2 weeks prior to enrollment;
3. Participant has severe co-morbidities that in the opinion of the investigator pose the patient at undue risk from participating in the study;
4. Participant has an active or past medical history of leptomeningeal disease;
5. Participant has spinal cord compression that has not been definitively treated with surgery or radiation or requires steroid treatment within 2 weeks prior to enrollment. Low-dose corticosteroid treatment ≤10mg/day prednisone or equivalent is allowed;
6. Participant has an active or past medical history of Interstitial lung disease (ILD)/pneumonitis, including drug-induced or radiation ILD/pneumonitis;
7. Immune-mediated rash from checkpoint inhibitors that has not resolved prior to enrollment;
8. Subject has uncontrolled inter-current illness;
9. Participant has active cardiovascular disease;
10. Participant is currently receiving medications or herbal supplements known to be potent CYP3A4/5 inhibitors or inducers and is unable to stop use for an appropriate washout period prior to enrollment (see Appendix 8: Prohibited and Restricted Medications and Therapies That Induce, Inhibit, or Are Substrates of CYP3A4/5);
11. Participant has received any prior treatment with an EGFR TKI;
12. Known positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg);
13. Known positive hepatitis C antibody (anti-HCV). Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible;
14. Other clinically active or chronic liver disease;
15. Known active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), Patients positive for human immunodeficiency virus (HIV) can be eligible if receiving highly active antiretroviral therapy (ART) and CD4 count >350 within 6 months of the start of treatment (consultation of Medical Monitor is required in this case). Screening for tuberculosis, hepatitis B, hepatitis C, and/or HIV infections is not required, unless there is clinical suspicion of these infections;
16. Participant had major surgery (e.g., requiring general anesthesia), excluding placement of vascular access or tumor biopsy, or had significant traumatic injury within 2 weeks before signing the ICF, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 18-month progression-free survival (PFS) rate | 18 months
  To evaluate the 18-month progression-free survival (PFS) rate of amivantamab, lazertinib, carboplatin and pemetrexed for first-line treatment of recurrent / metastatic non-small cell lung cancers (NSCLCs) with EGFR mutations.

SECONDARY OUTCOMES:
Overall progression-free survival | 18 months
Overall response rate | 18 months
  Defined as the proportion of complete response (CR) or partial response (PR) according to RECIST v1.1.
Overall survival | 18 months
  Overall survival is defined as the time from the date of enrollment to the date of participant's death due to any cause.
Progression-free survival After First Subsequent Therapy (PFS 2) | 18 months
  The PFS 2 is defined as the time from enrollment until the date of second objective disease progression, after initiation of subsequent anticancer therapy, based on investigator assessment (after that used for PFS) or death, whichever comes first.
Incidence of Treatment-Emergent Adverse Events and toxicity assessed by CTCAE v5.0 | 18 months
  Safety includes adverse events in terms of treatment-emergent adverse events (AE). The rate of any grade of adverse events as well as the rate of adverse events grade ≥3 according to the CTCAE version 5 will be evaluated. Adverse events of special interest of Amivantamab and Lazertinib will be based on the definitions given in the protocol of each one.
Performance status at progression-free survival 1 and progression-free survival 2 | 18 months
Compliance | 18 months
  Includes number of patients whose treatment had to be reduced, delayed, or permanently discontinued, grouped by reason. The reason for termination includes aspects of efficacy (e.g. termination due to tumor progression), safety (e.g. termination due to adverse events) and compliance (e.g. termination due to patient's withdrawal of consent).
Post-progression therapies | 18 months
  Description of therapies after disease progression.
Patient reported outcomes | 18 months
  Defined as the change from baseline of disease-related symptoms and quality of life based on European Organization for Research and Treatment of Cancer (EORTC) core cancer instrument and supplemental lung cancer module.
Intracranial Progression-Free Survival | 18 months
  Intracranial PFS is defined as the time from enrollment until the date of objective intracranial disease progression or death, whichever comes first, using RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: William Nassib William Junior, Principal Investigator — Latin American Cooperative Oncology Group
Locations (14):
- Brazil (14):
  - Pronutrir - Oncologia e Nutrição, Fortaleza, Ceará
  - Hospital Evangélico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - Centro de Tratamento de Tumores Botafogo (Oncoclínicas), Rio de Janeiro
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - São Camilo Oncologia, São Paulo